CLINICAL TRIAL: NCT05921565
Title: Mobile - PrOmoting Wellness After cancER Study: M-POWER Feasibility Study
Brief Title: M-POWER Feasibility Study
Acronym: M-POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Professor of Preventive Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00207968
Record Dates: First submitted 2023-05-15; First posted 2023-06-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Weight Reduction; Adherence, Patient
MeSH Terms: conditions — Weight Loss; Patient Compliance

STUDY DESIGN:
Intervention Model Description: To explore individual differences in responses to the weight loss intervention as well as mechanisms underlying its effects, additional survey measures will be administered. These measures will include: demographics, other health information, motivations for losing weight (TSR-Q), personality (BFI-10), chronic stress (Life Events Inventory) perceived stress (PSS-10), stress in past week, the positive and negative affect scale, PROMIS scale of cognitive function PROMIS scales of physical function, PROMIS scales of mental health, PROMIS scales of social health, fear of cancer recurrence, and self-efficacy for diet and exercise. PROMIS items will be assessed using computerized adaptive testing versions with items drawn from banks specific to the individual constructs assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Behavioral Arm (Experimental): Everyone in the study will receive the same type of treatment. They will all receive a treatment period that will last for 8 weeks. All participants will be given a 3% total weight loss goal, a daily calorie goal ranging from 1200-2000 kcal/day based on body weight, and a daily fat goal based on 25% of total daily calories from fat, and an option to stop their food/energy intake at 6pm every day without altering any other meal times. .Participants will also be asked to use two meal replacements per day. Participants will also be given a physical activity goal of 100 minutes per week.
  Interventions: Behavioral: Interventional Behavioral Arm

INTERVENTIONS:
Behavioral: Interventional Behavioral Arm — All participants will receive a weight loss intervention that includes 8 coaching sessions guided by a workbook they will at their baseline visit. During these sessions, they will meet with a health coach individually for up to 10-15 minutes via telephone or video conference to learn and discuss weight loss strategies. Health coaches will provide feedback and instruction (by phone or email) based on progress and challenges encountered during the intervention. Participants will receive a weight management app custom-built for the research study. The app will display participants' dietary intake, physical activity, and weight data and goals on the smartphone, and participants will use the app to log dietary intake, physical activity, and weight daily.

SUMMARY:
The purpose of this study is to test a new weight loss intervention designed for cancer survivors who have heart disease or cardiometabolic conditions. The investigators want to determine whether this study is feasible and acceptable to participants. The investigators also want to learn more about how cancer survivors take their medications.

DETAILED DESCRIPTION:
The purpose of this study is to test a new weight loss intervention designed for cancer survivors. The investigators want to determine whether this approach to weight loss is feasible and acceptable to cancer survivors. All participants in the study will receive free behavioral telephone-based weight loss management in the Department of Preventive Medicine at Northwestern University. Participants must be willing and able to use their smartphone with Bluetooth and their WiFi to download Apps, set up a Fitbit account and a Google account if not already set up. Participants will use their smartphone to record food intake & physical activity over an 8 week weight loss program. This program includes recruitment of a "Buddy" that the participant will choose to support you during the 8 week study.

All participants will be asked to download a study application to use to record dietary intake each day during a "Run-In Week.". Eligible participants will then receive an 8-week weight loss program, including individual weekly sessions with health coaches. The investigators will also ask participants to complete both a baseline and follow-up session with study staff. If permitted by current university policies, these sessions will be held at the offices on Northwestern University's Chicago campus. Otherwise, these sessions will be conducted remotely via Zoom videoconference. If this is the case, as a privacy safeguard, the waiting room feature will be applied so that study staff can control who is admitted into the meeting. We expect that the participants will be in this research study for about 10 weeks.

The primary risk of participation is muscle soreness or injury from increased physical activity, as well as feelings of hunger from making changes to diet. The main benefit is that a participant may experience positive changes to their health and mood based on the study.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors between ages 18 and 84
* BMI between ≥25 - 45 kg/m2
* <350 lbs.; weight stable (no loss or gain >15 lbs. for the past 3 months)
* Own a smartphone (Android or iOS) and web camera, be willing to install the M-POWER App
* Will voluntarily provide informed consent
* Reside in the Chicagoland area for the duration of their participation (i.e., 3 months)
* Maintain at-home internet and WiFi service for the entirety of their participation
* Cancer survivors with a history of breast cancer (up to stage IIIa), melanoma (up to stage IIb), prostate cancer (up to stage IIIb) or colorectal cancer (up to stage IIIa).

Exclusion Criteria:

* Inability to speak and read English
* Unstable medical conditions

  * Uncontrolled hypertension
  * Diabetes - uncontrolled or treated with insulin
  * Uncontrolled hypothyroidism
  * Unstable angina pectoris
  * Transient ischemic attack
  * Cancer undergoing active treatment (< 3 months since most recent surgery, chemotherapy, or radiation treatment for cancer)
  * Cerebrovascular accident or myocardial infarction within the past six months, Crohn's disease)
  * Pregnancy, lactation or intended pregnancy
  * Active suicidal ideation
  * Anorexia
  * Bulimia
  * Binge eating disorder
  * Requiring an assistive device for mobility, or those with any current condition that may limit or prevent participation in moderate physical activity
  * Upcoming reconstructive surgery scheduled to take place during the study period and/or < 3months have elapsed since reconstructive surgery
  * Substance abuse or dependence besides nicotine dependence
  * Active treatment of the primary cancer
  * Individuals that have ever had bariatric (or LapBand surgery)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - Weight - Aria Scale | Baseline (week one) & Follow Up (week 8)
  Weight will be measured in the lab at baseline and then the change in weight at the follow-up. Baseline measurements occur one week before the study and follow up measurements occur at week 8 of the study. Measurements will be taken without shoes, wearing light clothing on a calibrated beam balance scale called the Aria Scale.
  For melanoma patients only, skin self-examination frequency will also be assessed.

SECONDARY OUTCOMES:
Additional Physiologic Outcomes | Baseline (week one) & Follow Up (week 8)
  Height will also be measured using a stadiometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States